CLINICAL TRIAL: NCT06697470
Title: Cross-sectional Study on the Variation of Muscle Thickness and Subcutaneous Tissues by Ultrasound and Bioelectrical Impedance in Association with the Fluid Balance of Patients in Intensive Care
Brief Title: Muscle and Subcutaneous Tissue Variation by Ultrasound and Impedance Linked to Fluid Balance in ICU Patients
Status: Recruiting | Type: Observational
Sponsor: Dr F Duprez (Other)
Responsible Party: Sponsor-Investigator, Dr F Duprez, Physiotherapist / Professor at Provincial High School Condorcet (PhD) & Director of the Unité de recherche et d'innovation Condorcet EpiCURA (URICE), Laboratory of Movement, Condorcet, Tournai, Belgium
Organization: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Other Study IDs: P2024/372
Record Dates: First submitted 2024-10-28; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Weakness Acquired in the ICU; Muscle Wasting; Edema; Fluid Overload; Critical Illness; Intensive Care Unit (ICU) Patients
Keywords: Muscle thickness; Subcutaneous tissue; Ultrasound; Bioelectrical impedance analysis; BIA; Fluid balance; ICU (intensive care unit); Muscle strength; MRC-sum score; Grip strength; Edema assessment; Critical care; Skeletal muscle; Hydration status; Muscle echogenicity; ICU-acquired weakness; Fluid compartments; Extracellular water; Intracellular water; Body composition; Bedside ultrasound; Fluid management; Early mobilization; Volume overload; Tissue edema; Body water compartments; Length of ICU stay; Muscle quality
MeSH Terms: conditions — Muscular Atrophy; Edema; Critical Illness | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically Ill Patients in ICU: This cohort consists of adult patients aged over 18 years who are admitted to the ICU at Epicura Hornu Hospital between October 14, 2024, and November 15, 2024 (to be updated). The study will investigate muscle thickness variations and fluid balance using ultrasound and bioelectrical impedance analysis (BIA). Informed consent will be obtained from the patients or their legal representatives.
  Interventions: Device: Ultrasound and Bioelectrical Impedance Analysis for Muscle Thickness and Fluid Balance Assessment Translation

INTERVENTIONS:
Device: Ultrasound and Bioelectrical Impedance Analysis for Muscle Thickness and Fluid Balance Assessment Translation — This intervention involves the use of ultrasound and bioelectrical impedance analysis (BIA) to monitor changes in muscle thickness and assess fluid balance in critically ill patients. Measurements will be taken daily during the patients' ICU stay, with a focus on rectus femoris, tibialis anterior, and biceps brachii muscles, as well as total body fluid compartments. The study aims to explore correlations between muscle thickness variations, fluid balance, and patient outcomes.

SUMMARY:
This cross-sectional study aims to investigate the relationship between variations in muscle thickness and subcutaneous tissue, measured by ultrasound, and fluid compartments, evaluated using bioelectrical impedance analysis (BIA), in critically ill patients in the intensive care unit (ICU). Critically ill patients frequently experience muscle wasting and tissue edema due to a combination of inflammation, immobilization, and aggressive fluid resuscitation protocols designed to counteract hemodynamic instability.

Ultrasound is widely used to monitor muscle thickness because it is fast, non-invasive, and repeatable. However, muscle thickness measurements during the first days of ICU admission may be influenced by fluid overload, which causes edema and might lead to an overestimation of actual muscle mass. Bioelectrical impedance analysis (BIA) is a complementary tool that assesses both intra- and extracellular fluid compartments. This study aims to correlate daily fluid balance with changes in muscle thickness and subcutaneous tissue measured by ultrasound, and to determine if BIA can accurately reflect fluid status and potentially identify edema in these patients.

Furthermore, at ICU discharge, patients' muscle strength will be assessed using both the MRC-sum score (0-60) and handgrip strength (using a Jamar dynamometer), to investigate whether the presence of edema at discharge correlates with muscle strength deficits. Data collection will occur daily, tracking fluid balance, clinical parameters, and body weight, alongside ultrasound and BIA measurements in a standardized position. The study will help clarify the interactions between fluid management, muscle mass changes, and clinical outcomes in critically ill patients, providing valuable insight into early rehabilitation strategies.

DETAILED DESCRIPTION:
Muscle wasting and edema are common complications in critically ill patients, particularly those requiring intensive care. The rapid decrease in muscle mass and strength, known as ICU-acquired weakness, affects both peripheral and respiratory muscles, reducing patients' functional capacity in both the short and long term. Early interventions like physical therapy and mobilization have been shown to improve patient outcomes, but there is a need for accurate monitoring of muscle mass and fluid balance during the ICU stay to guide treatment.

This study leverages two complementary measurement techniques: ultrasound and bioelectrical impedance analysis (BIA). Ultrasound allows for the rapid and non-invasive assessment of muscle thickness and subcutaneous tissues. Previous studies have demonstrated that patients in the ICU can lose around 2% of their rectus femoris muscle thickness per day during the first week of their ICU stay. Ultrasound can also assess the structural changes in muscle tissue, such as alterations in echogenicity, that occur due to the inflammatory state of critically ill patients. However, patients undergoing aggressive fluid resuscitation to counteract shock and hypotension may experience fluid overload, which can distort early ultrasound measurements by causing tissue edema.

Bioelectrical impedance analysis (BIA), on the other hand, is a widely used method for evaluating body composition, particularly in terms of fat-free mass, fat mass, and fluid compartments. In the ICU, BIA is highly sensitive to changes in fluid balance, providing estimates of extracellular and intracellular water. This makes BIA particularly useful for tracking fluid shifts and edema development over time in critically ill patients.

The primary objective of this study is to explore the correlation between daily fluid balance and the changes in muscle thickness and subcutaneous tissue, as measured by ultrasound, and to assess the utility of BIA in evaluating fluid status and estimating the presence of edema. Specifically, the study will address two main research questions: (1) Is there a correlation between fluid balance and muscle thickness or subcutaneous tissue variation during the ICU stay? (2) Can BIA accurately reflect positive fluid balance and help estimate the extent of tissue edema?

The study will also include an exploratory analysis at ICU discharge to determine whether there is a link between the presence of edema and patients' muscle strength. Muscle strength will be assessed using both the MRC-sum score (0-60) and handgrip strength with a Jamar dynamometer. Previous studies have shown that ICU-acquired weakness is associated with poorer long-term outcomes, and this study will explore whether edema contributes to this weakness.

Patients will be recruited according to predefined inclusion and exclusion criteria. Upon obtaining consent from the patient or their legal representative, baseline clinical data (age, sex, BMI, reason for ICU admission, comorbidities, and severity scores such as APACHE-2 and SOFA) will be collected. Daily data will include vital signs, ventilatory settings, fluid balance, body weight, and medication details. Ultrasound and BIA measurements will be taken daily, with the patient positioned in a standardized way (supine position with a 30° incline). The ultrasound measurements will focus on the rectus femoris, tibialis anterior, and biceps brachii muscles, along with key subcutaneous tissues prone to fluid accumulation. BIA measurements will estimate total body water, extracellular water (ECW), intracellular water (ICW), muscle mass, and fat mass.

At ICU discharge, handgrip strength and MRC-sum score measurements will be performed to assess functional recovery and muscle strength. This study will provide valuable insights into how fluid management and edema contribute to muscle wasting and weakness in critically ill patients, informing future therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years.
* Patients present and admitted to the ICU at Epicura Hornu Hospital between October 14, 2024, and November 15, 2024 (to be updated).
* Informed consent to participate in the study has been signed by the patient or their legal representative.

Exclusion Criteria :

* Patients in post-operative or other surveillance with an expected ICU stay of less than 48 hours.
* Patients for whom a decision to withdraw therapy has been made prior to inclusion.
* Presence of skin conditions (e.g., wounds or ulcers) that hinder ultrasound measurements or the application of skin electrodes.
* Pregnancy.
* Presence of an implanted pacemaker or defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of critically ill adult patients aged over 18 years, admitted to the Intensive Care Unit (ICU) at the Centre Hospitalier Epicura Hornu between October 14, 2024, and November 15, 2024 (to be updated). Participants will include individuals who have provided informed consent to participate in the study or whose legal representatives have signed on their behalf. The cohort will represent a diverse range of medical conditions requiring intensive care, and all participants will be monitored for muscle thickness variation and fluid balance throughout their ICU stay.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness Variation Measured by Ultrasound (US) | Daily from the date of ICU admission until ICU discharge or up to a maximum of 28 days.
  Daily change in muscle thickness assessed by ultrasound (e.g., rectus femoris, tibialis anterior, and biceps brachii) from ICU admission to discharge. Muscle thickness will be measured in millimeters (mm) to evaluate muscle loss during the ICU stay.
  Unit of Measure: Millimeters (mm)
Fluid Balance Using Bioelectrical Impedance Analysis (BIA) | Daily from the date of ICU admission until ICU discharge or up to a maximum of 28 days.
  Daily change in total body water, extracellular water, and intracellular water assessed by bioelectrical impedance analysis (BIA) from ICU admission to discharge. Fluid compartments will be measured in liters (L), and the values will provide insights into fluid balance and its relationship to muscle changes during critical illness.
  Unit of Measure: Liters (L)

SECONDARY OUTCOMES:
Grip Strength Assessment | Grip strength will be assessed once at the time of ICU discharge, which is expected to occur within 2 to 28 days of ICU admission.
  This outcome measure evaluates grip strength using a dynamometer (Jamar hand dynamometer) at the time of ICU discharge. Grip strength will be assessed in the dominant hand, with three repetitions recorded to determine the maximum strength output. This measure will provide insights into the functional status and muscular strength of patients as they transition out of the ICU.
  Unit of Measure:
  Pounds (lb)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Epicura site Hornu, Boussu, Hainaut
  - Epicura site Hornu, Boussu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gonzalez-Seguel F, Pinto-Concha JJ, Rios-Castro F, Silva-Gutierrez A, Camus-Molina A, Mayer KP, Parry SM. Evaluating a Muscle Ultrasound Education Program: Theoretical Knowledge, Hands-on Skills, Reliability, and Satisfaction of Critical Care Physiotherapists. Arch Rehabil Res Clin Transl. 2021 Jul 13;3(3):100142. doi: 10.1016/j.arrct.2021.100142. eCollection 2021 Sep. PMID 34589692
- [Background] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Background] Grimm A, Teschner U, Porzelius C, Ludewig K, Zielske J, Witte OW, Brunkhorst FM, Axer H. Muscle ultrasound for early assessment of critical illness neuromyopathy in severe sepsis. Crit Care. 2013 Oct 7;17(5):R227. doi: 10.1186/cc13050. PMID 24499688
- [Background] Formenti P, Umbrello M, Coppola S, Froio S, Chiumello D. Clinical review: peripheral muscular ultrasound in the ICU. Ann Intensive Care. 2019 May 17;9(1):57. doi: 10.1186/s13613-019-0531-x. PMID 31101987
- [Background] Malbrain ML, Huygh J, Dabrowski W, De Waele JJ, Staelens A, Wauters J. The use of bio-electrical impedance analysis (BIA) to guide fluid management, resuscitation and deresuscitation in critically ill patients: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):381-91. doi: 10.5603/AIT.2014.0061. PMID 25432557
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Manuel Gomez J, Lilienthal Heitmann B, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, M W J Schols A, Pichard C; ESPEN. Bioelectrical impedance analysis-part II: utilization in clinical practice. Clin Nutr. 2004 Dec;23(6):1430-53. doi: 10.1016/j.clnu.2004.09.012. PMID 15556267
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Reynolds PM, Stefanos S, MacLaren R. Restrictive resuscitation in patients with sepsis and mortality: A systematic review and meta-analysis with trial sequential analysis. Pharmacotherapy. 2023 Feb;43(2):104-114. doi: 10.1002/phar.2764. Epub 2023 Jan 21. PMID 36625778
- [Background] Murphy CV, Schramm GE, Doherty JA, Reichley RM, Gajic O, Afessa B, Micek ST, Kollef MH. The importance of fluid management in acute lung injury secondary to septic shock. Chest. 2009 Jul;136(1):102-109. doi: 10.1378/chest.08-2706. Epub 2009 Mar 24. PMID 19318675
- [Background] Fazzini B, Markl T, Costas C, Blobner M, Schaller SJ, Prowle J, Puthucheary Z, Wackerhage H. The rate and assessment of muscle wasting during critical illness: a systematic review and meta-analysis. Crit Care. 2023 Jan 3;27(1):2. doi: 10.1186/s13054-022-04253-0. PMID 36597123
- [Background] Paolo F, Valentina G, Silvia C, Tommaso P, Elena C, Martin D, Marini John J, Davide C. The possible predictive value of muscle ultrasound in the diagnosis of ICUAW in long-term critically ill patients. J Crit Care. 2022 Oct;71:154104. doi: 10.1016/j.jcrc.2022.154104. Epub 2022 Jul 4. PMID 35797827
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Parry SM, Puthucheary ZA. The impact of extended bed rest on the musculoskeletal system in the critical care environment. Extrem Physiol Med. 2015 Oct 9;4:16. doi: 10.1186/s13728-015-0036-7. eCollection 2015. PMID 26457181
- [Background] Latronico N, Rasulo FA, Eikermann M, Piva S. Illness Weakness, Polyneuropathy and Myopathy: Diagnosis, treatment, and long-term outcomes. Crit Care. 2023 Nov 13;27(1):439. doi: 10.1186/s13054-023-04676-3. PMID 37957759